CLINICAL TRIAL: NCT05372939
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group, Exploratory, Phase 2 Study of the Efficacy and Safety of Oral AMT-101 in Combination With Adalimumab in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Study of the Efficacy and Safety of AMT-101 in Combination With Adalimumab in Subjects With Ulcerative Colitis (MARKET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Applied Molecular Transport (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMT-101-203
Record Dates: First submitted 2021-09-22; First posted 2022-05-13 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMT-101 and Humira (adalimumab) (Active Comparator): AMT-101 Tablet
  Interventions: Drug: AMT-101 (oral); Combination Product: Humira (adalimumab)
- Placebo and Humira (adalimumab) (Placebo Comparator): Placebo Tablet
  Interventions: Other: Placebo (oral); Combination Product: Humira (adalimumab)

INTERVENTIONS:
Drug: AMT-101 (oral) — AMT 101 is orally administered biological therapeutic taken once daily
  Arms: AMT-101 and Humira (adalimumab)
Other: Placebo (oral) — Orally administered placebo comparator taken once daily
  Arms: Placebo and Humira (adalimumab)
Combination Product: Humira (adalimumab) — Humira comparator is administered subcutaneously, on Humira frequency schedule.

SUMMARY:
Randomized, Placebo-controlled, Double-blind, Parallel-group, Multicenter, Phase 2a Study of the Efficacy and Safety of Oral AMT-101 in Combination With Adalimumab in Subjects with Moderate to Severe Ulcerative Colitis.

DETAILED DESCRIPTION:
This is a Randomized, Placebo-controlled, Double-blind, Parallel-group, Multicenter, Phase 2a Study to evaluate the Efficacy and Safety of Oral AMT-101 in Combination with Adalimumab in Subjects with Moderate to Severe Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 75 years.
* Moderate to severe UC.
* Eligible for Humira (adalimumab) therapy.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening and at the randomization visit.
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* Known gastrologic, or systemic condition that may compromise severity or diagnosis of disease.
* History or current evidence of colonic or abdominal abnormalities.
* Prohibited therapies or procedures before the screening period as specified per protocol.
* A concurrent clinically significant, serious, unstable, or uncontrolled underlying cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, might confound the study results, pose additional risk to the subject, or interfere with the subject's ability to participate fully in the study.
* Pregnant or lactating females.
* Current or recent history of alcohol dependence, illicit drug use, mental or legal incapacitation, or a history of clinically significant psychiatric disorders that, in the opinion of the investigator, may interfere with the subject's ability to comply with the study procedures.
* Unable to attend study visits or comply with procedures.
* Previous exposure to AMT-101 or similar and known hypersensitivity to AMT-101 or its excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Ulcerative Colitis disease activity as assessed by mean change in UC-100 Score from baseline | 8 weeks
  To evaluate the effects of AMT-101 in combination with adalimumab on ulcerative colitis (UC) disease activity

SECONDARY OUTCOMES:
Mean change in Robarts Histopathology Index (RHI) from baseline | 8 weeks
Mean change in total Mayo Clinic Score (MCS) and component scores (Mayo Endoscopic Subscore [MES], partial MCS, rectal bleeding and stool frequency) from baseline | 8 weeks
Mean change in fecal calprotectin from baseline | 8 weeks
Mean change in high-sensitivity C-reactive protein (hs-CRP) from baseline | 8 weeks
Proportion of subjects who achieve a significant reduction in RHI | 8 weeks
Clinical remission rate | 8 weeks
Clinical response rate | 8 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Arensia Exploratory Medicine GmbH Georgia, Tbilisi, Georgia
- Academic Medical Center, Amsterdam, Netherlands
- Poland (10):
  - NZOZ Vitamed, Bydgoszcz
  - Centrum Medyczne LukaMed Joanna Łuka-Wendrowska, Chojnice
  - Centrum Medyczne CLW-med Aneta Cichomska , Joanna Łuka -Wendrowska, Grudziądz
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Centrum Innowacyjnych Terapii Sp. z o.o. Oddzial w Piasecznie, Piaseczno
  - Centrum Medyczne Medyk, Rzeszów
  - H.T. Centrum Medyczne - Endoterapia, Tychy
  - Niepubliczny Zakład Opieki Zdrowotnej Vivamed Jadwiga Miecz, Warsaw
  - Bodyclinic sp z o.o. Sp. Kom., Warsaw
  - Centrum Medyczne Melita Medical, Wroclaw
- Ukraine (6):
  - Medical Center of Limited Liability Company "Harmoniya Krasy", Kyiv
  - Medical Center "OK!Clinic+" of International Institute of Clinical Research LLC, Gastroenterology and Hepatology unit of Hospital department, Kyiv
  - Municipal non-profit enterprise of Kyiv Regional Council "Kyiv Regional Hospital", Therapeutic Department, Kyiv
  - Municipal non-profit enterprise "Vinnytsia Regional Clinical Hospital named after M.I. Pirogov of Vinnytsia Regional Council", Regional Specialized Clinical gastroenterological Center, Vinnytsia
  - Municipal non-profit enterprise "Vinnytsya City Clinical Hospital No1", Gastroenterology Department, Vinnytsia
  - Medical Center of Limited Liability Company "Medibor", Department of Daycare, Day Surgery with Intensive Care Ward, Zhytomyr